CLINICAL TRIAL: NCT06661317
Title: Presence of HIV-1 DRMs As a Risk Factor of Failure of Two Drugs Based ART Regimens, Including LAI ART, in Cohorts of Primary and Secondary DRMs.
Brief Title: Primary and Secondary Drug Resistance Mutations (DRMs) in HIV As a Risk Factor of Failure of ART, Including Two Drugs Based Regimens.
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: Primary and secondary HIV DRMs
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-06

CONDITIONS: HIV-1-infection; DRM; DRM Gene Mutation; ART
Keywords: HIV; drug resistance mutations; DRM; LAI; ART; integrase inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- primary DRMs: patients with the presence of primary DRMs
  Interventions: Other: no intervention
- secondary DRMs: patients with the presence of secondary DRMs
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The presence of drug resistance mutations (DRMs) in HIV plays an important role in ART effectiveness. Despite very good results of ART, there is constant concern about the emergence of HIV strains with DRMs, what may lead to virological suppression failure. The concerns grow especially among patients treated with two drugs based regimens, including long acting therapies in injections (LAI ART) or regimens used in preexposure prophylaxis (PreP).

DETAILED DESCRIPTION:
Introduction The presence of drug resistance mutations (DRMs) in HIV plays an important role in ART effectiveness. Despite very good results of ART, there is constant concern about the emergence of HIV strains with DRMs, what may lead to virological suppression failure. Primary HIV DRMs occur in PLWH who have not previously been treated with ART. These people start treatment with a lower genetic barrier, a higher risk of virological failure and a higher risk of developing resistance to other drugs, which may lead to progression to AIDS. The concerns grow especially among patients treated with two drugs based regimens, including long acting therapies in injections (LAI ART) or regimens used in preexposure prophylaxis (PreP). The prevalence of major HIV-1 DRMs reported worldwide ranges from 5 to 25%, while in case of accessory (polymorphic) DRMs even up to 50%. It has been reported that in high-income countries the prevalence of sequences with acquired DRMs is decreasing, but the fraction of transmitted resistance is clearly increasing compared to the fraction of acquired DRMs, reaching even 70% of all cases of DRMs.

Aim of the study The choice of ART is based on epidemiological data regarding the presence of drug resistance mutations in HIV, as well on the basis of the HIV genotyping test results assessed before the start or change of the treatment. The presence of DRMs before ART initiation may be a risk factor for insufficient virological suppression, as the population of HIV is still evolving (changing due to mistakes during replication process). As well, inadequate antiretroviral therapy may drive the viral population first through a lower fitness level and then to a higher fitness level. Due to the constant changes in the pattern of HIV drug resistance (emergence of new mutations) and the introduction of new drugs into the treatment, including two drugs based regimens as LAI ART, we decided to conduct a study which determine the type and frequency of DRMs (including NRTI and NNRTI - RPV, 3TC and InSTI - CAB, DTG), in the population of previously untreated patients, as well as among patients with ART virological failure. The results may help in assessing the risk of ART failure, including LAI, and in determining ART regimens.

Methodology We aim to conduct multi-center, observational, cross sectional study. The patients' data will be extracted from the 2 year period (2023 - 2024). The site of the recruitment will be three clinical centers in Poland (two in Warsaw, one in Ostróda). Inclusion criteria are: diagnosis with HIV-1 infection, age 18 years or older. We will collect epidemiological data such as: age, gender, BMI, route of transmission also clinical and laboratory findings: HIV viral load, lymphocyte CD4 count and CD4:CD8 ratio (at the time of diagnosis/ change of therapy), presence of AIDS-defining diseases, implemented ART regimen. In all patients, before starting ART, the presence of HIV-1 DRMs to nucleoside reverse transcriptase inhibitors (NRTI), non-nucleoside reverse transcriptase inhibitors (NNRTI) protease inhibitors (PI) and integrase inhibitors (InSTI) will be evaluated, as a part of routine care.

The drug resistance genotyping of HIV-1 protease (PR) and reverse transcriptase (RT) coding region will be performed based on a Sanger sequencing method with use of commercially available ViroSeq HIV-1 Genotyping System (Abbott Molecular, Des Plains, IL, USA). The analysis procedure will be performed according to the manufacturer's instructions. HIV-1 RNA will be extracted manually from 0,5 mL of collected plasma samples by precipitation and centrifugation steps, followed by reverse transcription with MuLV reverse transcriptase. DNA products corresponding to the 1.8 kb pol region fragment will be generated in PCR with AmpliTaq Gold DNA Polymerase, after pre-incubation with Uracil-N-Glycosylase (UNG) enzyme. Where HIV-1 integrase coding region will be sequenced the ViroSeq HIV-1 Integrase Genotyping System (Celera Diagnostics, Alameda, CA, USA) will be applied with one step RT-PCR amplification reaction. Obtained PCR products will be purified enzymatically by incubation with Exo-SAP mix (Exonuclease I + Shrimp Alkaline Phosphatase), diluted if necessary, fluorescently labelled in reaction with appropriate terminators and sequenced by ABI Prism 3130 Genetic Analyzer using Data Collection Software (Applied Biosystems). The resulting sequence chromatograms will be assembled and analyzed using ViroSeq Genotyping System Software (Abbott Molecular). Drug resistance-associated mutations in protease, integrase and reverse transcriptase will be identified. The valid, quality checked pol sequences will be submitted to the Stanford University HIV Drug Resistance Database (http://hivdb.stanford.edu) in order to comparison of potential differences in the interpretation of the significance of genetic variants detected. For HIV-1 subtype and circular recombinant forms (CRFs) determination of partial pol submitted sequences REGA HIV-1 Subtyping Tool Version 3.0 will be used.

Statistical evaluation of the collected data will be performed in subgroups of PLWH with the presence of primary and secondary HIV DRMs. The analysis will also be performed in the subgroups of patients with different subtype HIV-1 infection. The Shapiro-Wilk test will be performed for the verification of the normality of the distributions in the analyzed variables. Student's t-test or Mann-Whitney U test will be used to evaluate the difference in mean value in continuous variables and χ 2 or Fisher exact tests will be performed for categorical variables. A p value of <0.05 will be considered statistically significant. Statistical analyses will be performed using Python 3.7 software and Statistica 13.1 program (StatSoft Poland, Kraków, Poland).

The clinical trial has received a positive opinion from the Bioethics Committee at the Medical University of Warsaw (number of consent: AKBE/72/2023). All analyzed patients' data will be fully anonymized. The study follows the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were: diagnosis with HIV-1 infection, age 18 years or older.

Exclusion Criteria:

Lack of HIV genotyping before ART treatment or change of ART

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV- 1 diagnosed patient recruited in three clinical centers in Poland (two in Warsaw, one in Ostróda)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
frequency of DRMs | 2 years
  frequency of DRMs in all included patients

SECONDARY OUTCOMES:
frequency of primary and secondary DRMs | 2 years
  frequency of primary and secondary DRMs, including resistance to InSTI

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Załęski, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Infectious Diseases, Tropical Diseases and Hepatology, Medical University of Warsaw, Warsaw, Mazowia, Poland

IPD SHARING:
Plan to Share IPD: No
data extracted from medical records

REFERENCES:
- [Background] Rhee SY, Kassaye SG, Barrow G, Sundaramurthi JC, Jordan MR, Shafer RW. HIV-1 transmitted drug resistance surveillance: shifting trends in study design and prevalence estimates. J Int AIDS Soc. 2020 Sep;23(9):e25611. doi: 10.1002/jia2.25611. PMID 32936523
- [Background] Wensing AM, Calvez V, Ceccherini-Silberstein F, Charpentier C, Gunthard HF, Paredes R, Shafer RW, Richman DD. 2022 update of the drug resistance mutations in HIV-1. Top Antivir Med. 2022 Oct;30(4):559-574. PMID 36375130
- [Background] Mazzuti L, Melengu T, Falasca F, Calabretto M, Cella E, Ciccozzi M, Mezzaroma I, Iaiani G, Spaziante M, d'Ettorre G, Fimiani C, Vullo V, Antonelli G, Turriziani O. Transmitted drug resistance mutations and trends of HIV-1 subtypes in treatment-naive patients: A single-centre experience. J Glob Antimicrob Resist. 2020 Mar;20:298-303. doi: 10.1016/j.jgar.2019.08.024. Epub 2019 Sep 10. PMID 31518723
- [Background] Swindells S, Lutz T, Van Zyl L, Porteiro N, Stoll M, Mitha E, Shon A, Benn P, Huang JO, Harrington CM, Hove K, Ford SL, Talarico CL, Chounta V, Crauwels H, Van Solingen-Ristea R, Vanveggel S, Margolis DA, Smith KY, Vandermeulen K, Spreen WR. Week 96 extension results of a Phase 3 study evaluating long-acting cabotegravir with rilpivirine for HIV-1 treatment. AIDS. 2022 Feb 1;36(2):185-194. doi: 10.1097/QAD.0000000000003025. PMID 34261093
- [Background] Landovitz RJ, Donnell D, Clement ME, Hanscom B, Cottle L, Coelho L, Cabello R, Chariyalertsak S, Dunne EF, Frank I, Gallardo-Cartagena JA, Gaur AH, Gonzales P, Tran HV, Hinojosa JC, Kallas EG, Kelley CF, Losso MH, Madruga JV, Middelkoop K, Phanuphak N, Santos B, Sued O, Valencia Huamani J, Overton ET, Swaminathan S, Del Rio C, Gulick RM, Richardson P, Sullivan P, Piwowar-Manning E, Marzinke M, Hendrix C, Li M, Wang Z, Marrazzo J, Daar E, Asmelash A, Brown TT, Anderson P, Eshleman SH, Bryan M, Blanchette C, Lucas J, Psaros C, Safren S, Sugarman J, Scott H, Eron JJ, Fields SD, Sista ND, Gomez-Feliciano K, Jennings A, Kofron RM, Holtz TH, Shin K, Rooney JF, Smith KY, Spreen W, Margolis D, Rinehart A, Adeyeye A, Cohen MS, McCauley M, Grinsztejn B; HPTN 083 Study Team. Cabotegravir for HIV Prevention in Cisgender Men and Transgender Women. N Engl J Med. 2021 Aug 12;385(7):595-608. doi: 10.1056/NEJMoa2101016. PMID 34379922
- [Background] Bokharaei-Salim F, Esghaei M, Khanaliha K, Kalantari S, Marjani A, Fakhim A, Keyvani H. HIV-1 reverse transcriptase and protease mutations for drug-resistance detection among treatment-experienced and naive HIV-infected individuals. PLoS One. 2020 Mar 2;15(3):e0229275. doi: 10.1371/journal.pone.0229275. eCollection 2020. PMID 32119691
- [Background] Richardson D, Fitzpatrick C, Parkes L, Roberts J, Mulka L. HIV-1 transmitted drug resistance in Brighton, UK, from 2014 to 2020. Int J STD AIDS. 2021 Feb;32(2):199-201. doi: 10.1177/0956462420953043. Epub 2020 Dec 16. PMID 33327896
- [Background] Branda F, Giovanetti M, Sernicola L, Farcomeni S, Ciccozzi M, Borsetti A. Comprehensive Analysis of HIV-1 Integrase Resistance-Related Mutations in African Countries. Pathogens. 2024 Jan 24;13(2):102. doi: 10.3390/pathogens13020102. PMID 38392840
- [Background] Scherrer AU, von Wyl V, Yang WL, Kouyos RD, Boni J, Yerly S, Klimkait T, Aubert V, Cavassini M, Battegay M, Furrer H, Calmy A, Vernazza P, Bernasconi E, Gunthard HF; Swiss HIV Cohort Study; Aubert V, Battegay M, Bernasconi E, Boni J, Braun DL, Bucher HC, Burton-Jeangros C, Calmy A, Cavassini M, Dollenmaier G, Egger M, Elzi L, Fehr J, Fellay J, Furrer H, Fux CA, Gorgievski M, Gunthard H, Haerry D, Hasse B, Hirsch HH, Hoffmann M, Hosli I, Kahlert C, Kaiser L, Keiser O, Klimkait T, Kouyos R, Kovari H, Ledergerber B, Martinetti G, Martinez de Tejada B, Marzolini C, Metzner K, Muller N, Nadal D, Nicca D, Pantaleo G, Rauch A, Regenass S, Rudin C, Schoni-Affolter F, Schmid P, Speck R, Stockle M, Tarr P, Trkola A, Vernazza P, Weber R, Yerly S. Emergence of Acquired HIV-1 Drug Resistance Almost Stopped in Switzerland: A 15-Year Prospective Cohort Analysis. Clin Infect Dis. 2016 May 15;62(10):1310-1317. doi: 10.1093/cid/ciw128. Epub 2016 Mar 8. PMID 26962075
- [Background] Rossetti B, Di Giambenedetto S, Torti C, Postorino MC, Punzi G, Saladini F, Gennari W, Borghi V, Monno L, Pignataro AR, Polilli E, Colafigli M, Poggi A, Tini S, Zazzi M, De Luca A; Antiviral Response Cohort Analysis (ARCA) Collaborative Group. Evolution of transmitted HIV-1 drug resistance and viral subtypes circulation in Italy from 2006 to 2016. HIV Med. 2018 Oct;19(9):619-628. doi: 10.1111/hiv.12640. Epub 2018 Jun 22. PMID 29932313
- [Background] Pingarilho M, Pimentel V, Diogo I, Fernandes S, Miranda M, Pineda-Pena A, Libin P, Theys K, Martins MRO, Vandamme AM, Camacho R, Gomes P, Abecasis A. Increasing Prevalence of HIV-1 Transmitted Drug Resistance in Portugal: Implications for First Line Treatment Recommendations. Viruses. 2020 Oct 30;12(11):1238. doi: 10.3390/v12111238. PMID 33143301
- [Background] Nijhuis M, Schuurman R, de Jong D, Erickson J, Gustchina E, Albert J, Schipper P, Gulnik S, Boucher CA. Increased fitness of drug resistant HIV-1 protease as a result of acquisition of compensatory mutations during suboptimal therapy. AIDS. 1999 Dec 3;13(17):2349-59. doi: 10.1097/00002030-199912030-00006. PMID 10597776